CLINICAL TRIAL: NCT01385891
Title: Clofarabine, Cyclophosfamide, And Etoposide For The Treatment Of Relapsed Or Resistant Acute Leukemia In Pediatric Patients
Brief Title: Clove In The Treatment Of Relapsed Or Resistant Acute Leukemia In Children
Acronym: CLOVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: lorenzo moretta, G Gaslini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM001; 2008-004487-39 (EudraCT Number)
Record Dates: First submitted 2011-06-21; First posted 2011-06-30 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Acute Leukemia
MeSH Terms: interventions — Clofarabine; Etoposide; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- children with advanced leukemia (Experimental)
  Interventions: Drug: Clofarabine VP 16 ciclophospahamide

INTERVENTIONS:
Drug: Clofarabine VP 16 ciclophospahamide — Clofarabine intravenously 2-hour infusion,dose 40 mg/m2, followed by Etoposide (VP 16)100 mg/m2 i.v. over 2 hours and Cyclophosphamide 440 mg/m2 i.v. over 1 hour
  Other Names: Evoltra; Etoposide; Endoxan

SUMMARY:
Study Hypothesis. combination chemotherapy with Clofarabine VP16 and Cyclophosphamide is able to induce remission in resistant/refractory acute leukemias in pediatric.

Forty children with relapsed or refractory Acute Lymphoblastic Leukemia (ALL) or Acute Myeloid Leukemia (AML) entered the study and received the association of clofarabine (40 mg/m2/day) in combination with etoposide (100 mg/m2/day) and Cyclophosphamide (440 mg/m2/day) in 1 or 2 induction cycles End point were complete remission (CR)or CR without platelet recovery (CRp) and toxicity

ELIGIBILITY:
Inclusion Criteria:

* presence of > 25% of blast in bone marrow
* treatment with second line therapies
* patients with resistant disease i.e. with >25% of blasts 21 days after the last cytostatic agent administration
* children with persistent high MRD level (> 10-3) after first or further line chemotherapy, were considered eligible to the treatment
* Relapsed after > months after SCT
* Karnofsky score >50
* a Forced Espiratory Volume >30%
* sufficient hepatic and renal function defined as creatinine levels <2 × ULN, bilirubin <1.5 × ULN
* aspartate and alanine aminotransferases <10 × ULN.

Exclusion Criteria:

* isolated extra-medullary relapse, and active infections

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
response to treatment | after an expected average of 3 weeks after the first dose of each chemotherapy course

SECONDARY OUTCOMES:
Number of patients with toxicity as a measure of safety and tolerability | at an expected average of 4 weeks after the first dose of each chemotherapy course
  Grade of toxicity defined according to the National Cancer's Inst. Common terminology Criteria (NCI CTCAE v3.0)

CONTACTS AND LOCATIONS:
Overall Officials: Concetta Micalizzi, MD, Principal Investigator — G. Gaslini Hospital
Locations (1):
- G.Gaslini Children's Hospital, Genova, Italy